CLINICAL TRIAL: NCT03580655
Title: An Open-label, Single Arm, Phase 2 Study to Evaluate Efficacy and Safety of Avapritinib (BLU-285), A Selective KIT Mutation-targeted Tyrosine Kinase Inhibitor, in Patients With Advanced Systemic Mastocytosis
Brief Title: (PATHFINDER) Study to Evaluate Efficacy and Safety of Avapritinib (BLU-285), A Selective KIT Mutation-targeted Tyrosine Kinase Inhibitor, in Patients With Advanced Systemic Mastocytosis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Blueprint Medicines Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BLU-285-2202; 2017-004836-13 (EudraCT Number)
Record Dates: First submitted 2018-05-03; First posted 2018-07-09 (Actual); Last update posted 2025-04-30 (Actual); Status verified 2025-04

CONDITIONS: Advanced Systemic Mastocytosis; Aggressive Systemic Mastocytosis; Systemic Mastocytosis With an Associated Hematologic Neoplasm; Mast Cell Leukemia
MeSH Terms: conditions — Mastocytosis, Systemic; Leukemia, Mast-Cell | interventions — avapritinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Avapritinib (Experimental): Avapritinib will be administered as an immediate release tablet, orally, continuously, in 28-day cycles
  Interventions: Drug: Avapritinib

INTERVENTIONS:
Drug: Avapritinib — Avapritinib tablet
  Other Names: BLU-285

SUMMARY:
This is an open-label, single arm, Phase 2 study evaluating the efficacy and safety of avapritinib (BLU-285) in patients with advanced systemic mastocytosis (AdvSM), including patients with aggressive SM (ASM), SM with associated hematologic neoplasm (SM-AHN), and mast cell leukemia (MCL)

ELIGIBILITY:
Key Inclusion Criteria:

1. Patient must have a diagnosis of aggressive systemic mastocytosis (ASM), systemic mastocytosis with an associated hematologic neoplasm (SM-AHN) or mast cell leukemia (MCL) based on World Health Organization diagnostic criteria. Before enrollment, the Study Steering Committee must confirm the diagnosis of AdvSM (based on Central Pathology Laboratory assessment of bone marrow).
2. Patient must have a serum tryptase ≥ 20 ng/mL.
3. Patient must have Eastern Cooperative Oncology Group (ECOG) performance status (PS) of 0 to 3.

Key Exclusion Criteria:

1. Patient has received prior treatment with avapritinib.
2. Patient has received any cytoreductive therapy (including midostaurin and other TKIs, hydroxyurea, azacitidine) or an investigational agent less than 14 days, and for cladribine, interferon alpha, pegylated interferon and any antibody therapy (eg, brentuximab vedotin) less than 28 days before obtaining screening BM biopsy for this study.
3. Patient has eosinophilia and known positivity for the FIP1L1 PGDFRA fusion, unless the patient has demonstrated relapse or PD on prior imatinib therapy. Patients with eosinophilia (> 1.5 × 10^9/L), who do not have a detectable KIT D816 mutation, must be tested for a PDGFRA fusion mutation by fluorescence in situ hybridization (FISH) or polymerase chain reaction (PCR).
4. Patient has history of another primary malignancy that has been diagnosed or required therapy within 3 years before the first dose of study drug. The following are exempt from the 3-year limit: completely resected basal cell and squamous cell skin cancer, curatively treated localized prostate cancer, and completely resected carcinoma in situ of any site.
5. Patient has a QT interval corrected using Fridericia's formula (QTcF) > 480 msec.
6. Patient has a known risk or recent history (12 months before the first dose of study drug) of intracranial bleeding (eg, brain aneurysm, concomitant vitamin K antagonist use).
7. Platelet count < 50,000/μL (within 4 weeks of the first dose of study drug) or receiving platelet transfusion(s).
8. Aspartate aminotransferase (AST) or alanine aminotransferase (ALT) >3 x the upper limit of normal (ULN); no restriction if due to suspected liver infiltration by mast cells.
9. Bilirubin >1.5 × ULN; no restriction if due to suspected liver infiltration by mast cells or Gilbert's disease. (In the case of Gilbert's disease, a direct bilirubin >2 × ULN would be an exclusion.)
10. Estimated glomerular filtration rate (eGFR) < 30 mL/min/1.73m2 or creatinine > 1.5 × ULN.
11. Patient has a primary brain malignancy or metastases to the brain.
12. Patient has a history of a seizure disorder (eg, epilepsy) or requirement for antiseizure medication.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 107 (Actual)
Dates: Start 2018-11-21 (Actual); Primary Completion 2024-12-18 (Actual); Study Completion 2024-12-18 (Actual)

PRIMARY OUTCOMES:
Objective response rate (ORR) based on modified International Working Group-Myeloproliferative Neoplasms Research and Treatment and European Competence Network on Mastocytosis (IWG-MRT-ECNM) response criteria | 10 Months

SECONDARY OUTCOMES:
Mean Change from Baseline in Advanced Systemic Mastocytosis-Symptom Assessment Form (AdvSM-SAF) Total Symptom Score | 10 Months
  0 - 80 points (higher value represents worse symptom outcomes)
Objective response rate | Approximately 4 years after the first subjected enrolled
  Including morphologic complete remission (mCR), morphologic CR with partial recovery of peripheral blood (mCRh), and morphologic partial remission (mPR) based on Pure Pathologic Response
Time-to-response (TTR) | 10 Months
  Months
Duration of Response (DOR) | 10 Months
  Months
Progression-free Survival (PFS) | 10 Months
  Months
Overall Survival (OS) | 10 Months
  Months
Changes in bone marrow mast cells | 10 Months
  percentage
Change in serum tryptase | 10 Months
  ng/mL
Change in V-kit Hardy-Zuckerman 4 feline sarcoma viral oncogene homolog aspartate 816 valine (KIT D816V) mutation burden | 10 Months
  percentage
Change in liver volume by imaging | 10 Months
  mL
Change in spleen volume by imaging | 10 Months
  mL
Clinical benefit based on modified IWG-MRT-ECNM consensus criteria | 10 Months
Change in PGIS | 10 Months
  0 - 10 points (higher value represents worse symptom outcomes)
Change in EORTC QLQ-C30 | 10 Months
  0 - 100 points (lower value represents worse quality of life)
Safety of Avapritinib as assessed by incidence of adverse events | 10 Months
  CTCAE version 4.0
Area Under Curve (0 to Tau) for Avapritinib | 4 Months
  h•ng/mL

CONTACTS AND LOCATIONS:
Locations (32):
- United States (12):
  - Stanford Cancer Institute, Stanford, California
  - Rush University Medical Center, Chicago, Illinois
  - The University of Kansas Cancer Center, Westwood, Kansas
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - University of Michigan, Ann Arbor, Michigan
  - Washington University School of Medicine, St Louis, Missouri
  - Roswell Park Comprehensive Cancer Center, Buffalo, New York
  - Herbert Irving Comprehensive Cancer Center, New York, New York
  - University of Pennsylvania, Abramson Cancer Center, Philadelphia, Pennsylvania
  - University of Texas, MD Anderson Cancer Center, Houston, Texas
  - Mays Cancer Center, San Antonio, Texas
  - Huntsman Cancer Institute, Salt Lake City, Utah
- Medizinische Universität Wien, Universitätsklinik für Innere Medizin I, Klinische Abteilung für Hämatologie und Hämostaseologie, Vienna, Austria
- St. Michael's Hospital, Toronto, Ontario, Canada
- Odense University Hospital, Department of Haematology, Odense, Denmark
- France (2):
  - Hôpital Necker-Enfants Malades, Paris
  - CHU Toulouse - Hôpital Larrey, Toulouse
- Germany (5):
  - Uniklinik RWTH Aachen, Klinik für Hämatologie, Onkologie, Hämostaseologie und Stammzelltranslplantation, Aachen
  - Universitätsklinikum Hamburg-Eppendorf, Zentrum für Onkologie, Hamburg
  - Universitätsklinikum Leipzig, Medizinische Klinik und Poliklinik I - Hämatologie und Zelltherapie, lnternistische Onkologie, Hämostaseologie, Leipzig
  - Universitätsmedizin Mannheim III. Medizinische Klinik, Mannheim
  - Klinik und Poliklinik für Innere Medizin III, Klinikum rechts der Isar der TU München, Munich
- Italy (3):
  - Azienda Ospedaliero-Universitaria Careggi, CRIMM - Centro di Ricerca ed Innovazione per le Malattie Mieloproliferative, Florence
  - A.O. OO.RR. S.Giovanni di Dio e Ruggi d'Aragona, University of Salerno, Salerno
  - Centro Ricerche Cliniche di Verona - Azienda Ospedaliera Universitaria Integrata di Verona, Verona
- University Medical Center Groningen (UMCG), Groningen, Netherlands
- Oslo University Hospital-Rikshospitalet, Hematology, Oslo, Norway
- Poland (2):
  - Uniwersyteckie Centrum Kliniczne, Klinika Hematologii i Transplantologii, Gdansk
  - Uniwersytecki Szpital Kliniczny im. Jana Mikulicza-Radeckiego we Wrocławiu, Klinice Hematologii, Nowotworów Krwi i Transplantacji Szpiku, Wroclaw
- lnstituto de Estudios de Mastocitosis de Castilla la Mancha, Hospital Virgen del Valle - Complejo Hospitalario de Toledo, Toledo, Spain
- United Kingdom (2):
  - Beatson West of Scotland Cancer Centre - NHS Greater Glasgow and Clyde, Glasgow
  - Guy's and St Thomas' NHS Foundation Trust - Guy's Hospital, London

REFERENCES:
- [Derived] Reiter A, Gotlib J, Alvarez-Twose I, Radia DH, Lubke J, Bobbili PJ, Wang A, Norregaard C, Dimitrijevic S, Sullivan E, Louie-Gao M, Schwaab J, Galinsky IA, Perkins C, Sperr WR, Sriskandarajah P, Chin A, Sendhil SR, Duh MS, Valent P, DeAngelo DJ. Efficacy of avapritinib versus best available therapy in the treatment of advanced systemic mastocytosis. Leukemia. 2022 Aug;36(8):2108-2120. doi: 10.1038/s41375-022-01615-z. Epub 2022 Jul 5. PMID 35790816
- [Derived] Reiter A, Schwaab J, DeAngelo DJ, Gotlib J, Deininger MW, Pettit KM, Alvarez-Twose I, Vannucchi AM, Panse J, Platzbecker U, Hermine O, Dybedal I, Lin HM, Rylova SN, Ehlert K, Dimitrijevic S, Radia DH. Efficacy and safety of avapritinib in previously treated patients with advanced systemic mastocytosis. Blood Adv. 2022 Nov 8;6(21):5750-5762. doi: 10.1182/bloodadvances.2022007539. PMID 35640224
- [Derived] Gotlib J, Reiter A, Radia DH, Deininger MW, George TI, Panse J, Vannucchi AM, Platzbecker U, Alvarez-Twose I, Mital A, Hermine O, Dybedal I, Hexner EO, Hicks LK, Span L, Mesa R, Bose P, Pettit KM, Heaney ML, Oh ST, Sen J, Lin HM, Mar BG, DeAngelo DJ. Efficacy and safety of avapritinib in advanced systemic mastocytosis: interim analysis of the phase 2 PATHFINDER trial. Nat Med. 2021 Dec;27(12):2192-2199. doi: 10.1038/s41591-021-01539-8. Epub 2021 Dec 6. PMID 34873345